CLINICAL TRIAL: NCT06720831
Title: Role of Mesh in Laparoscopic Sacropexy Surgical Techniques for the Treatment of Female Genital Prolapse
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SACROMESH
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Female Genital Prolapse
Keywords: prolapse; female genital; gynaecology; sacropexy; mesh
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to determine the rate of recurrence of central pelvic organ prolapse in patients who have undergone surgery (sacropexy with and without mesh) for the same pathology.

DETAILED DESCRIPTION:
There is a lack of data in the literature comparing sacroplexing with the use of mesh with sacroplexing performed without the use of mesh in terms of recurrence, improvement in symptoms, and restoration of normal pelvic organ prolapse relationships. The objective of this study is to determine the rate of recurrence of central pelvic organ prolapse in patients with a clinical diagnosis of genital prolapse stage ≥ 2 according to the POP-Q classification who underwent laparoscopic sacroplasty with mesh (group 1) and without mesh (group 2). The study may provide information on the impact of mesh in laparoscopic surgery for the correction of central pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of genital prolapse stage ≥ 2 according to POP-Q classification
* Surgical treatment of laparoscopic sacropexy by mesh (group 1) and without (group 2) in female patients
* Acquisition of informed consent
* At least one follow-up evaluation at 24 months

Exclusion Criteria:

* Age > 80 years
* Previous genital prolapse surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with genital prolapse stage ≥ 2 according to the POP-Q classification undergoing laparoscopic sacroplexxy with mesh and laparoscopic sacropexy without mesh
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of central pelvic organ prolapse | 24 months after surgery
  The rate of recurrence of central pelvic organ prolapse in patients with a clinical diagnosis of genital prolapse stage ≥ 2 according to the POP-Q classification, undergoing sacroplasty with and without mesh

SECONDARY OUTCOMES:
Recurrence rate of central pelvic organ prolapse in laparoscopic sacral hysteropexy, sacralcervicopexy and sacralcolpopexy | 24 months after surgery
  The rate of pelvic organ prolapse recurrence in patients treated with mesh (group 1) and without (group 2) in the laparoscopic sacral hysteropexy, sacralcervicopexy and sacralcolpopexy
Rate of intraoperative and postoperative complications | During surgery and within 30 days
  Evaluation of intraoperative and postoperative complications according to the Clavien-Dindo classification
Modification of symptoms after surgery | Before surgery and 24 months after surgery
  Change in pre- and post-operative symptomatology assessed through the completion of a questionnaire
Changes in the disease framework | Before surgery and 24 months after surgery
  Change in the disease framework of pelvic organ prolapse according to the POP-Q classification assessed before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Verona